CLINICAL TRIAL: NCT02712099
Title: TUI 3D in Diagnosis of Placenta Accreta: Comparison With Gray-scale and Color Doppler Techniques
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rehab Mohamed Abdelrahman, Lecturer of Obstetrics and Gynaecology Faculty of Medicine, Ain Shams University, Ain Shams University
Other Study IDs: TUI 3D
Record Dates: First submitted 2016-03-09; First posted 2016-03-18 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate the potential of the 3 D TUI view in diagnosis of morbidly adherent placenta in comparison to 2D grayscale, color Doppler and intraoperative findings.

DETAILED DESCRIPTION:
* This is a prospective study which will include 50 patients who will be selected from the outpatient and inpatient obstetric Ain Shams university maternity hospital.
* All patients will undergo the following :

  1. History taking
  2. Clinical examination.
  3. For each patient, the whole placenta will be scanned in a systematic fashion using both 2D grayscale and 2D power Doppler ultrasound then displayed by 3D TUI to determine whether those patients suspected of having advanced invasive placentation.

ELIGIBILITY:
Inclusion Criteria:

1. History of previous cesarean section or hysterotomy.
2. Placenta previa with its lower edge covering the scar of previous cesarean section
3. From 28 wks to Full term.

Exclusion Criteria:

1. Multiple pregnancies.
2. Medical disorder as diabetes mellitus, hypertension.
3. Obese patients. BMI > 30
4. Intrauterine growth retardation.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * This is a prospective study which will include 50 patients who will be selected from the outpatient and inpatient obstetric Ain Shams university maternity hospital.
  * All patients will undergo the following :
    1. History taking
    2. Clinical examination.
    3. For each patient, the whole placenta will be scanned in a systematic fashion using both 2D grayscale and 2D power Doppler ultrasound then displayed by 3D TUI to determine whether those patients suspected of having advanced invasive placentation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
TUI 3D in Diagnosis of Placenta Accreta: Comparison with Gray-scale and Color Doppler Techniques
  * This is a prospective study which will include 50 patients who will be selected from the outpatient and inpatient obstetric Ain Shams university maternity hospital.
  * Patient consent should be taken first.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: study that was performed at the Fetal Care Unit at Ain Shams University Maternity Hospital from August 2015 to march 2016.
  Fifty pregnant women In whom the transabdominal scan revealed evidence of anterior placenta previa were recruited from the the Fetal Care Unit who fulfilled the inclusion criteria.
Groups:
- Women With Placenta Previa Who Had Easily Placenta Delivery: This is a prospective study which will include 50 patients who will be selected from the outpatient and inpatient obstetric Ain Shams university maternity hospital.
  • All patients will undergo the following : For each patient, the whole placenta will be scanned in a systematic fashion using both 2D grayscale and 2D power Doppler ultrasound then displayed by 3D TUI to determine whether those patients suspected of having advanced invasive placentation.
  Intraoperative:
  * Delivery of the fetus through the placenta.
  * 15 minutes for spontaneous separation of the placenta were waited, if easily separated hot packs then rapid closure of the uterus in 2 layers.
    30 Women with placenta previa who had easily placenta delivery
- Women With Placenta Previa Who Had Difficult Placenta Delivery: This is a prospective study which will include 50 patients who will be selected from the outpatient and inpatient obstetric Ain Shams university maternity hospital.
  • All patients will undergo the following : For each patient, the whole placenta will be scanned in a systematic fashion using both 2D grayscale and 2D power Doppler ultrasound then displayed by 3D TUI to determine whether those patients suspected of having advanced invasive placentation.
  Intraoperative:
  * Delivery of the fetus through the placenta.
  * 15 minutes for spontaneous separation of the placenta were waited, if easily separated hot packs then rapid closure of the uterus in 2 layers.
  * When not separated easily manual removal was done, with uterotonics, together with uterine massage.
    20 Women with placenta previa who had difficult placenta delivery
Period: Overall Study
Arm/Group | Women With Placenta Previa Who Had Easily Placenta Delivery | Women With Placenta Previa Who Had Difficult Placenta Delivery
Started | 30 | 20
Completed | 30 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Fifty pregnant women In whom the transabdominal scan revealed evidence of anterior placenta previa were recruited from the the Fetal Care Unit who fulfilled the inclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Women With Placenta Previa Who Had Easily Placenta Delivery | Women With Placenta Previa Who Had Difficult Placenta Delivery | Total
Number analyzed (Participants) | 30 | 20 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 20 | 50
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 20 | 50
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Egypt | 30 | 20 | 50

OUTCOME MEASURES:

1. Primary Outcome: Loss of the Retro Placental Sonolucent Zone by 2D Grayscale Ultrasonography
Description: 2D grayscale ultrasonography criteria of placenta accreta by Loss of the retro placental sonolucent zone in placenta previa with its lower edge covering the scar of previous cesarean section
Time Frame: 28 -36 weeks of gestation
Measure: Number; unit: participants
Arm/Group | Women With Placenta Previa Who Had Easily Placenta Delivery | Women With Placenta Previa Who Had Difficult Placenta Delivery
Number analyzed (Participants) | 30 | 20
participants | 12 | 19

2. Primary Outcome: Abnormal Placental Lacunae by 2D Grayscale Ultrasonography
Description: 2D grayscale ultrasonography criteria of placenta accreta by Abnormal placental lacunae in placenta previa with its lower edge covering the scar of previous cesarean section
Time Frame: 28 -36 weeks of gestation
Measure: Number; unit: participants
Arm/Group | Women With Placenta Previa Who Had Easily Placenta Delivery | Women With Placenta Previa Who Had Difficult Placenta Delivery
Number analyzed (Participants) | 30 | 20
participants | 19 | 15

3. Secondary Outcome: Crowded Vessels Over Peripheral Sub-placental Zone by Power Doppler Ultrasonography
Description: Power Doppler ultrasonography criteria of Crowded vessels over peripheral sub-placental zone of in placenta previa with its lower edge covering the scar of previous cesarean section
Time Frame: 28 -36 weeks of gestation
Measure: Number; unit: participants
Arm/Group | Women With Placenta Previa Who Had Easily Placenta Delivery | Women With Placenta Previa Who Had Difficult Placenta Delivery
Number analyzed (Participants) | 30 | 20
participants | 8 | 18

4. Secondary Outcome: Abnormal Placental Lacunae by Power Doppler Ultrasonography
Description: Power Doppler ultrasonography criteria by Abnormal placental lacunae in placenta previa with its lower edge covering the scar of previous cesarean section
Time Frame: 28 -36 weeks of gestation
Measure: Number; unit: participants
Arm/Group | Women With Placenta Previa Who Had Easily Placenta Delivery | Women With Placenta Previa Who Had Difficult Placenta Delivery
Number analyzed (Participants) | 30 | 20
participants | 20 | 13

5. Secondary Outcome: Crowded Vessels Over Peripheral Sub-placental Zone by 3D Tomographic Ultrasound Imaging (TUI)
Description: the examiner can simultaneously display, on the monitor or on a hard copy, up to 24 preselected parallel cuts from a volume. The slices can be generated either along the initial or any other reconstructed plane of the region of interest (ROI) in intervals of 0.5 - to 5 mm segments. Slice thickness will be adjusted as necessary for each individual case. The most informative image among the multiple images will be displayed with the use of CrossXBeam, a postprocessing tool that allows one to enhance tissue and border differentiation, leading to sharper depiction of the tissue margins
Time Frame: 28 -36 weeks of gestation
Measure: Number; unit: participants
Arm/Group | Women With Placenta Previa Who Had Easily Placenta Delivery | Women With Placenta Previa Who Had Difficult Placenta Delivery
Number analyzed (Participants) | 30 | 20
participants | 7 | 18

6. Secondary Outcome: Abnormal Placental Lacunae by 3D Tomographic Ultrasound Imaging (TUI)
Description: 3D tomographic ultrasound imaging (TUI) of placenta previa with its lower edge covering the scar of previous cesarean section the examiner can simultaneously display, on the monitor or on a hard copy, up to 24 preselected parallel cuts from a volume. The slices can be generated either along the initial or any other reconstructed plane of the region of interest (ROI) in intervals of 0.5 - to 5 mm segments. Slice thickness will be adjusted as necessary for each individual case. The most informative image among the multiple images will be displayed with the use of CrossXBeam, a postprocessing tool that allows one to enhance tissue and border differentiation, leading to sharper depiction of the tissue margins
Time Frame: 28 -36 weeks of gestation
Measure: Number; unit: participants
Arm/Group | Women With Placenta Previa Who Had Easily Placenta Delivery | Women With Placenta Previa Who Had Difficult Placenta Delivery
Number analyzed (Participants) | 30 | 20
participants | 19 | 13

ADVERSE EVENTS:
Time Frame: from 28 weeks to 36 weeks of gestation
Description: Adverse Events were assessed during ultrasound examination
Arm/Group | Women With Placenta Previa Who Had Easily Placenta Delivery | Women With Placenta Previa Who Had Difficult Placenta Delivery
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/20
Other Adverse Events (participants affected / at risk) | 0/30 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No